CLINICAL TRIAL: NCT03078309
Title: A Controlled Study of the Effect of Cannabis on Visual Functions in Healthy Subjects and in Retinitis Pigmentosa Patients
Brief Title: The Effects of Cannabis on Visual Functions in Healthy and Retinitis Pigmentosa Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Hadas MECHOULAM, senior physician, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0007-17-HMO
Record Dates: First submitted 2017-02-10; First posted 2017-03-13 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Retinitis Pigmentosa; Retinal Degeneration; Cannabis
Keywords: retinitis pigmentosa; retinal degeneration; cannabis; THC; CBD; electrophysiology; visual functions; eye; retina
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Degeneration; Marijuana Abuse | interventions — nabiximols; Cannabidiol; Dronabinol

STUDY DESIGN:
Intervention Model Description: Arm 1 - healthy subjects. Arm 2 - subjects with retinitis pigmentosa All subjects will undergo a full ocular exam and visual functions will be assessed before and after the administration of a single dose of cannabis (THC:CBD 1:40). On the second study day all subjects will receive a single dose of cannabis (THC:CBD 1:1) and undergo the full ocular exam again.
Who Masked: Outcomes Assessor
Masking Description: Electrophysiology will be analyzed by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy (Experimental): All subjects will undergo a full ocular exam and visual functions will be assessed before and after the administration of a single dose of cannabis (THC:CBD 1:40). On the second study day all subjects will receive a single dose of cannabis (THC:CBD 1:1) and undergo the full ocular exam again.
  Interventions: Drug: cannabis
- Retinitis Pigmentosa (Experimental): All subjects will undergo a full ocular exam and visual functions will be assessed before and after the administration of a single dose of cannabis (THC:CBD 1:40). On the second study day all subjects will receive a single dose of cannabis (THC:CBD 1:1) and undergo the full ocular exam again.
  Interventions: Drug: cannabis

INTERVENTIONS:
Drug: cannabis — single dose sublingual cannabis (THC:CBD 1:1, THC:CBD 1:40)
  Other Names: cannabidiol; THC

SUMMARY:
Medical Marijuana is used widely, and its effects on the visual system and the function of the retina have not been investigated thoroughly. Some evidence suggests that cannabinoids may be beneficial in certain degenerative diseases of the retina.

The purpose of the study is

1. To determine whether cannabis derivatives affect the visual functions in healthy adults
2. To examine the effect of cannabis derivatives on the retina of retinitis pigmentosa patients

DETAILED DESCRIPTION:
Twenty five healthy subjects and 25 retinitis pigmentosa patients will be recruited and will sign an informed consent form. An initial eye exam will include visual acuity and stereo vision, eye movements and eye movement recording, a full slit lamp eye exam, intra-ocular pressure measurement, visual field, OCT and electrophysiology. The subjects will receive a single sublingual dose of cannabis (THC:CBD 1:1, THC 5 mg, or THE:CBD 1:40, THC 5 mg), and will undergo the above examination again. Subjects will be monitored for 5 hours after the administration of cannabis.

ELIGIBILITY:
Inclusion Criteria:

* consenting adults
* generally healthy with or without retinitis pigmentosa

Exclusion Criteria:

* chronic or acute disease other than retinitis pigmentosa
* use of medication
* congestive heart failure
* recent use of illicit drugs (past month)
* history of drug dependency
* history of psychiatric disorder in subject or immediate relatives
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Electroretinogram (ERG) - acivity of the neural retina mixed cone-rod response, cone flicker, rod response | 3 hours
  microvolt
Electroretinogram (ERG) - acivity of the neural retina cone flicker latency | 3 hours
  milliseconds

SECONDARY OUTCOMES:
Visual acuity | 3 hours
  LogMAR ETDRS
Titmus stereo eye movements | 3 hours
  seconds of arc
Eye movements | 3 hours
  degrees/second
Intra ocular pressure | 3 hours
  mmHg
Macular thickness (OCT) | 3 hours
  micrometers

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Mechoulam, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lax P, Esquiva G, Altavilla C, Cuenca N. Neuroprotective effects of the cannabinoid agonist HU210 on retinal degeneration. Exp Eye Res. 2014 Mar;120:175-85. doi: 10.1016/j.exer.2014.01.019. Epub 2014 Feb 1. PMID 24495949
- [Background] Russo EB, Merzouki A, Mesa JM, Frey KA, Bach PJ. Cannabis improves night vision: a case study of dark adaptometry and scotopic sensitivity in kif smokers of the Rif mountains of northern Morocco. J Ethnopharmacol. 2004 Jul;93(1):99-104. doi: 10.1016/j.jep.2004.03.029. PMID 15182912
- [Background] Lyons CJ, Robson AG. Retinal Ganglion Cell Dysfunction in Regular Cannabis Users: Is the Evidence Strong Enough to Consider an Association? JAMA Ophthalmol. 2017 Jan 1;135(1):60-61. doi: 10.1001/jamaophthalmol.2016.4780. No abstract available. PMID 27930772